CLINICAL TRIAL: NCT06475248
Title: Influence of Osteopathic Intervention on Cervical Muscles in Tension Headaches in Women: Randomized Controlled Trial
Brief Title: Influence of Osteopathic Intervention on Cervical Muscles in Tension Headaches in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Investigator, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OST1_014
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Tension Headaches
Keywords: Tension headaches; Trapezius Stretching; sternocleidomastoid Stretching; Suboccipital Inhibition; Manual Therapy; Osteopathy; HIT-6
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Each volunteer selected in this group will complete a scale, in this case Hit-6, to collect data and evaluate the evolution.
  Then a placebo technique will be used, which consists of imitating the contacts of the techniques without compressing or pulling the tissue, lasted 6 minutes.
  This procedure will be repeated for two more sessions. One month after the first evaluation, the volunteers filled out the Hit-6 scale again.
  Interventions: Other: Placebo Technique
- Experimental Group (Experimental): After each volunteer completes the Hit-6 scale, one of the researchers will perform the "trapezius and sternocleidomastoid stretching techniques", and "suboccipital inhibition". The techniques performed will only be done once, lasted 6 minutes.
  This procedure will be repeated for two more sessions. One month after the first evaluation, the volunteers filled out the Hit-6 scale again.
  Interventions: Other: Stretching technique; Other: Inhibition of the suboccipital

INTERVENTIONS:
Other: Placebo Technique — For the technique performed in the control group, the researcher will come into contact with the volunteers' chests. This contact will be maintained for the same period of time as the experimental group (6 minutes).
  Arms: Control Group
Other: Stretching technique — "Stretching technique" for the upper trapezius and sternocleidomastoid: the volunteer will be in supine position on the couch, the researcher will perform the technique from the contralateral side of the muscle to be treated, the hand will contact the ipsilateral shoulder to stabilize, meanwhile, with the other hand, contact the upper trapezius and perform a rhythmic pull in contralateral rotation. This technique is performed bilaterally.
  Arms: Experimental Group
Other: Inhibition of the suboccipital — "Inhibition of the suboccipital": the participant is in the supine position, the researcher will position himself behind the patients head. In this technique, contacts will be made on the suboccipital area with the 2nd, 3rd and 4th fingers of both hands. Make a slight pull with your body backwards and wait that there is relaxation of muscular tensions.
  Arms: Experimental Group

SUMMARY:
This study aims to understand whether there is any relationship between the intervention on the trapezius, sternocleidomastoid and suboccipital muscles in patients with chronic tension headaches.

DETAILED DESCRIPTION:
It is expected to find an improvement in the symptoms and frequency of tension headaches.

In this study, the investigators intend to see the effects of trapezius and sternocleidomastoid "stretching techniques", and "suboccipital inhibition" on tension headaches. To collect data, volunteers were asked to fill out the Headache Impact Test (HIT-6).

ELIGIBILITY:
Inclusion Criteria:

* Tension headaches;
* Being over eighteen years of age;

Exclusion Criteria:

* Loss of mobility of cervical;
* Cervical and shoulder pain during episodes;
* Other headaches (migraine, cervicogenic headache...)
* Other interventions and/or pharmacological treatment a few days before the intervention;
* Epilepsy;
* Trauma.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 43 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-11 (Estimated)

PRIMARY OUTCOMES:
Change in the intensity and frequency of pain after the three treatment sessions; | One month after the first intervention
  The scale Hit-6 will be the instrument used to evaluate the level the intensity and frequency of tension headache. This instrument consists of six questions about the characteristics of headaches, with each question presenting five choices. The answers range from never to always. This data will be collected immediately before the first investigation and one month after the first evaluation, through the volunteers filling out the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior da Saúde do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Cumplido-Trasmonte C, Fernandez-Gonzalez P, Alguacil-Diego IM, Molina-Rueda F. Manual therapy in adults with tension-type headache: A systematic review. Neurologia (Engl Ed). 2021 Sep;36(7):537-547. doi: 10.1016/j.nrleng.2017.12.005. Epub 2020 Apr 7. PMID 34537167
- [Background] Lebedeva ER, Kobzeva NR, Gilev DV, Olesen J. The quality of diagnosis and management of migraine and tension-type headache in three social groups in Russia. Cephalalgia. 2017 Mar;37(3):225-235. doi: 10.1177/0333102416642603. Epub 2016 Jul 11. PMID 27053061
- [Background] Hartman, L. S. (2013). Handbook of osteopathic technique. Springer